CLINICAL TRIAL: NCT05714540
Title: The Effect of Oropharyngeal Pack Soaked With Ketamine or Magnesium Sulphate on Post Operative Sore Throat After Nasal Surgeries: Randomized Controlled Double Blind Study
Brief Title: Effect of Oropharyngeal Pack Soaked in Ketamine or Magnesium Sulphate on Post Operative Sore Throat After Nasal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Jehan Mohamed Mohamed Abdelghany, Jehan Mohammed Mohammed Abdelghany, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OPP in nasal surgery
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Sore-throat; Nasopharyngeal Pack; Nasal Surgery; Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Pharyngitis; Postoperative Nausea and Vomiting | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): The patients will receive 20 ml 0.9% saline soaked pharyngeal pack inserted in the posterior pharyngeal wall after induction of anesthesia and endotracheal intubation .
  Interventions: Drug: Ketamine Hydrochloride ,Magnesium sulphate and saline 0.9%
- ketamine group (Active Comparator): The patients will receive ketamine soaked 50 mg ketamine in 20 ml normal saline soaked pharyngeal pack inserted in the posterior pharyngeal wall after induction of anesthesia and ETT insertion
  Interventions: Drug: Ketamine Hydrochloride ,Magnesium sulphate and saline 0.9%
- Magnesium group (Active Comparator): The patients will receive 20 mg/kg magnesium sulfate soaked pharyngeal pack inserted in the posterior pharyngeal wall after induction of anesthesia and ETT
  Interventions: Drug: Ketamine Hydrochloride ,Magnesium sulphate and saline 0.9%

INTERVENTIONS:
Drug: Ketamine Hydrochloride ,Magnesium sulphate and saline 0.9% — The Effect of Oropharyngeal Pack Soaked with Ketamine or Magnesium Sulphate on Post Operative Sore Throat after Nasal Surgeries

SUMMARY:
The aim of this study is to compare the effect of ketamine or magnesium sulphate soaked throat pack on the incidence and severity of post operative sore throat as a primary outcome, post operative nausea and vomiting as a secondary outcome following elective nasal surgery under general anesthesia.

DETAILED DESCRIPTION:
Postoperative sore throat (POST) is defined as pain, discomfort, or irritation in the throat after general anesthesia and tracheal intubation that worsens with swallowing. Etiological factors playing a significant role in this anesthetic complication are: Size of the endotracheal tube, design and pressure of cuff, the use of nasogastric tubes, lubricants, muscle relaxants, duration of surgery, surgery in and around the oral cavity, trauma arising from laryngoscopy, and use of pharyngeal packs. Pharyngeal packs are commonly used during nasal surgeries to prevent aspiration, tracheal contamination and passage of blood into the stomach. They are disputed to increase the incidence of postoperative sore throat (POST), but surgery in and around the oral cavity necessitates them to soak blood and debris that result as consequence of surgery and decrease post operative nausea and vomiting. Nausea and vomiting are important postoperative complications in all surgical settings and more in nasal surgery due to the presence of blood in the stomach, pain and inflammation of the uvula and throat, and the occasional use of opioids for pain control are all contributing factors. Many interventions can be used to decrease incidence of POST. These include using smaller endotracheal tube size including video laryngoscopy in intubation process, limiting endotracheal cuff pressure and perioperative use of steroids (intravenous, topical or inhaled). Also pharyngeal packs soaked with agents with analgesic effect can be used to decrease post operative sore throat, nausea and vomiting. N methyl D aspartate (NMDA) receptors are present in the central nervous system and also in the peripheral nervous system . These receptors contribute in inflammatory pain. Ketamine and Magnesium sulphate are NMDA antagonist with antinociceptive and anti-inflammatory effect, which may be a possible mechanism in prevention of postoperative sore throat (POST).

ELIGIBILITY:
Inclusion Criteria:

* The study will include 90 adult patients of American Society of Anesthesiologists (ASA) physical status I and II, in the age group of 18 to 60 years of age, of either sex, who will be scheduled for elective nasal surgery (e.g. unilateral or bilateral functional endoscopic sinus surgery, sub mucousal resection, septorhinoplasty , polypectomy) under general anesthesia with endotracheal intubation, having a Mallampatti Grades of I and II and those who are willing to give informed consent.

Exclusion Criteria:

* History of recent respiratory tract infection or sore throat , anticipated difficult airway, known allergy to study drug, and preoperative use of analgesics such as non-steroidal anti-inflammatory drugs or opioids, Patients who required more than one attempt for tracheal intubation, or who will need tracheal intubation of <60 minutes or>300 minutes will be eliminated from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
post operative sore throat | 24 hours

SECONDARY OUTCOMES:
nausea and vomiting | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine beni Suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No